CLINICAL TRIAL: NCT00712205
Title: Asthma and Vitamin D (a Clinical Pilot Study)
Brief Title: Vitamin D for the Treatment of Severe Asthma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kantonsspital Baselland Bruderholz (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Albrecht Breitenbücher MD, Department of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KSBH-336-06
Record Dates: First submitted 2008-06-26; First posted 2008-07-09 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Asthma
Keywords: Asthma; Vitamin D
MeSH Terms: conditions — Asthma | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): 20 Patients with asthma in a crossover design
  Interventions: Drug: Placebo
- B (Active Comparator): 20 Patients with asthma in a crossover design
  Interventions: Drug: Placebo; Drug: Calcitriol

INTERVENTIONS:
Drug: Placebo — once daily 1mcg Placebo for 28days followed by crossover treatment
Drug: Calcitriol — once daily 1mcg Calcitriol / Placebo for 28days followed by crossover treatment
  Arms: B

SUMMARY:
The investigators want to test the hypothesis, that vitamin D3 improves pulmonary function and quality of life in patients with asthma relatively resistant to glucocorticoids.

DETAILED DESCRIPTION:
Glucocorticoids are the first-line antiinflammatory treatment for asthma. Their multiple inhibitory properties, including the inhibition of Th2 cytokine synthesis, are likely to contribute to clinical efficacy. Glucocorticoids also enhance IL-10 production in vitro by human CD4+ and CD8+ T cells, and glucocorticoid treatment induces the synthesis of IL-10 by airway cells in asthmatic patients. IL-10 is a potent antiinflammatory and immunosuppressive leading to profound inhibition of Th1 cell-mediated immunity. A proportion of asthmatic patients fails to benefit from oral glucocorticoid therapy and are thus denoted as having glucocorticoid-resistant (SR, derived from "steroid resistant") or insensitive asthma. It has been demonstrated that CD4+ T cells from SR asthma patients fail to induce IL-10 synthesis following in vitro stimulation in the presence of dexamethasone as compared with their glucocorticoid-sensitive counterparts (SS, derived from "steroid sensitive"), suggesting a link between induction of IL-10 synthesis and clinical efficacy of glucocorticoids. One potential source of IL-10 is Tregs, which control the function of effector T cells. Glucocorticoids enhance the production of IL-10 by polyclonally stimulated T cells and these cells inhibit IFN- production by human CD4+ T cells in an IL-10-dependent manner. In both mouse and human a combination of dexamethasone and calcitriol, the active form of vitamin D3, induced high numbers of IL-10-producing T cells that made negligible amounts of Th1 and Th2 cytokines.

Xystrakis et al. (57) showed that IL-10-secreting Tregs inhibit cytokine production by previously activated allergen-specific Th2 cells and that pretreating T cells with IL-10 or adding vitamin D3 to the cell cultures can reverse the defect and enhance IL-10 production by Tregs from asthmatic patients who were resistant to glucocorticoid therapy. These manipulations increase IL-10 production to levels comparable to those observed in patients who do respond well to therapy. IL-10 increases glucocorticoid receptor expression, and the authors proposed that this is the mechanism by which IL-10 overcomes the glucocorticoid-resistant patient defect in IL-10 synthesis. This strongly suggests that vitamin D3 could potentially increase the therapeutic response to glucocorticoids in SR patients.

We want to test the hypothesis, that vitamin D3 improves pulmonary function and quality of life in patients with asthma relatively resistant to glucocorticoids.

ELIGIBILITY:
Inclusion Criteria:

* 20 outpatients of either sex,
* ages ≥18 years, with a history of persistent asthma as defined by the American Thoracic Society (ATS) will be eligible for entry into the study.
* Additionally, patients must have been previously treated with ICS for at least 4 weeks at a stable dose equivalent to ≥400 ug/day beclomethasone dipropionate.
* Patients will be required to have a forced expiratory volume in 1 s (FEV1) between 40-85% of predicted normal before the use of an inhaled bronchodilator and to demonstrate at least one of the following:

  * an improvement in FEV1 ≥ 12% and ≥ 200 ml within 15-30 min after inhalation of salbutamol 200-400 ug;
  * airway hyperresponsiveness to methacholine causing a 20% decline in FEV1 (PC20 FEV1) at a concentration of < 16 mg/ml;
  * diurnal peak expiratory flow (PEF) variability of ≥ 15% during at least 3 of 7 days before randomization.

Exclusion Criteria:

* Patients with either an exacerbation of asthma or respiratory tract infection within 6 weeks or admission to a hospital for asthma within 6 weeks before the study will be excluded.
* Also patients will not be eligible if they had > 3 nights with awakenings due to asthma that required treatment with short-acting betamimetics or had 3 days when they required > or = 12 puffs/d short-acting betamimetics during the 7days before the randomization visits.
* Patients will also excluded if they use medications greater potency than inhaled steroid, e.g.not leukotriene inhibitors or anti-IgE (Xolair®).
* Patients with chronic obstructive pulmonary disease and current or former smokers of >10 pack-years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
the area under the 12-hour serial FEV1 curve relative to day-1 baseline (FEV1 AUCbl) and bronchial responsiveness to methacholine | 4 weeks

SECONDARY OUTCOMES:
daily morning and evening PEF, daily patient-rated asthma symptom scores, short-acting betamimetics use, nighttime awakenings due to asthma requiring short-acting betamimetics use and the fraction of the exhaled nitric oxide (FENO). | daily

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Breitenbuecher, MD, Principal Investigator — Kantonsspital Baselland Bruderholz
Locations (1):
- Department of Medicine, Bruderholz, Basel-Landschaft, Switzerland

REFERENCES:
- [Derived] Lloyd CM, Hessel EM. Functions of T cells in asthma: more than just T(H)2 cells. Nat Rev Immunol. 2010 Dec;10(12):838-48. doi: 10.1038/nri2870. Epub 2010 Nov 9. PMID 21060320